CLINICAL TRIAL: NCT02619253
Title: A Phase I/Ib, Open Label, Dose Finding Study to Evaluate Safety, Pharmacodynamics and Efficacy of Pembrolizumab (MK-3475) in Combination With Vorinostat in Patients With Advanced Renal or Urothelial Cell Carcinoma
Brief Title: Phase I/Ib Study of Pembrolizumab With Vorinostat for Patients With Advanced Renal or Urothelial Cell Carcinoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Nabil Adra (Other)
Responsible Party: Sponsor-Investigator, Nabil Adra, Assistant Professor of Clinical Medicine, Indiana University School of Medicine
Organization: Indiana University (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IUSCC-0551
Record Dates: First submitted 2015-11-16; First posted 2015-12-02 (Estimated); Results first posted 2024-11-18 (Actual); Last update posted 2024-11-18 (Actual); Status verified 2024-09

CONDITIONS: Renal Cell Carcinoma; Urinary Bladder Neoplasms
Keywords: Immunotherapy; Safety; Pharmacodynamics; Efficacy
MeSH Terms: conditions — Carcinoma, Renal Cell; Urinary Bladder Neoplasms | interventions — pembrolizumab; Vorinostat

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Dose Finding Cohort (Experimental): Estimate the Recommended Phase 2 Dose (RP2D) in patients with advanced renal and urothelial cell carcinoma patients. Patients will be treated with oral vorinostat every day for 14 days, and with pembrolizumab at the fixed dose of 200 mg IV. Each cycle is every 21 days. Two dose levels of vorinostat will be tested in 2 patient cohorts according to the 3 + 3 standard design (100 and 200 mg).
  Interventions: Drug: Pembrolizumab; Drug: Vorinostat
- Expansion Cohort (Experimental): Once the Expansion Test Dose is identified, the Dose Expansion Phase will be opened and the combination will be tested in patients with advanced renal cell or urothelial cell carcinoma. Forty-five patients with prior treatments will be enrolled in three expansion cohorts: 15 anti-PD1 naive renal and urothelial patients, 15 anti-PD1 resistant renal and urothelial patients (defined as patients with transient clinical response or without clinical response to prior immune-checkpoint inhibition), and 15 patients with androgen-sensitive or castration-resistant prostate cancer.
  Interventions: Drug: Pembrolizumab; Drug: Vorinostat

INTERVENTIONS:
Drug: Pembrolizumab
  Other Names: Keytruda
Drug: Vorinostat
  Other Names: Zolinza

SUMMARY:
Primary objective: To assess the early signals for anti-tumor activity (i.e. objective response rate, progression-free survival) of pembrolizumab in combination with vorinostat in patients with advanced prostate, renal or urothelial cell carcinoma.

Secondary objectives: (1) To evaluate the overall safety profile of pembrolizumab in combination with vorinostat; (2) To assess the safety and tolerability of pembrolizumab in combination with vorinostat in patients with advanced prostate, renal or urothelial cell carcinoma in order to select the recommended Phase 2 Dose (RP2D)

DETAILED DESCRIPTION:
This is a Phase I/Ib, open-label, safety, and pharmacodynamics study of pembrolizumab in combination with vorinostat in patients with advanced prostrate, renal or urothelial cell carcinoma. This clinical study will be composed of a Dose Finding Phase and an Expansion Phase. The Dose Finding Phase will estimate the Recommended Phase II Dose (RP2D) in patients with advanced renal and urothelial cell carcinoma patients. The Dose Finding Phase will lead to the identification of an Expansion Test Dose for pembrolizumab in combination with vorinostat. The Expansion Test Dose will be the Recommended Phase II Dose (RP2D) (i.e. the highest tested dose that is declared safe and tolerable by the Investigators and Sponsor). Patients will be treated with oral vorinostat every day for 14 days, and with pembrolizumab at the fixed dose of 200 mg IV. Each cycle is every 21 days. Two dose levels of vorinostat will be tested in 2-patient cohorts according to the 3 + 3 standard design (100 mg and 200 mg). 200 mg dose represents 50% of the recommended vorinostat dose as single agent.

For the Dose Finding Phase (Combination Phase), the starting dose level of vorinostat will be 100 mg by mouth (PO) every day for 14 days, with 7 days break. The first dose level will have a minimum of 3 patients treated (unless the first 2 patients experience dose-limiting toxicities (DLTs) before the 3rd patient is enrolled).

Once the RP2D is identified, the Dose Expansion Phase will be opened. During the Dose Expansion Phase, the study will have a run-in phase with sequential single-agents and then the combination phase. The run-in phase may be waived at the investigator's discretion. The reason for the run-in phase during dose expansion is to obtain data on the immunomodulatory effects of vorinostat separately from pembrolizumab. Forty-five patients with prior treatments will be enrolled in three expansion cohorts: 15 anti-PD1 naive renal and urothelial patients 15 anti-PD1 resistant renal and urothelial patients (defined as patients with transient clinical response or without clinical response to prior immune-checkpoint inhibition), and 15 patients with androgen-sensitive or castration-resistant prostate cancer. The prostate cohort has been added in an amendment during the Dose Expansion Phase, and therefore, will not be part of the Dose Finding Phase.

ELIGIBILITY:
Subject Inclusion Criteria

In order to be eligible for participation in this trial, the subject must:

1. Have one of the following diagnoses/conditions:

   1. Renal cell carcinoma - previously treated and progressive disease, locally advanced or metastatic
   2. Urothelial cell carcinoma - previously treated and progressive disease, locally advanced or metastatic
   3. Prostate cell carcinoma - progressive disease, locally advanced or metastatic disease (enrolling only at IUSCC and its affiliates). Patients with hormone-sensitive disease where ADT in combination with either docetaxel or abiraterone is indicated will not be eligible (i.e. patients with high burden disease).
2. Be willing and able to provide written informed consent for the trial.
3. Be 18 years of age or older on day of signing informed consent.
4. Have measurable disease based on RECIST 1.1. for patients with solid malignancies or evaluable disease as assessed by bone scan and/or PET scan. Patients with advanced or metastatic prostate cancer can have either androgen-sensitive or castration-resistant disease.
5. Have a performance status of 0-2 on the ECOG Performance Scale.
6. Demonstrate adequate organ function. All screening labs should be performed within 10 days of treatment initiation.
7. Female subject of childbearing potential should have a negative urine or serum pregnancy test within 72 hours prior to receiving the first dose of study medication. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required.
8. Subjects of childbearing potential should be willing to use 2 methods of contraception for the course of the study through 120 days after the last dose of study medication. Acceptable methods of birth control include: abstinence, partner with previous vasectomy, placement of an intrauterine device (IUD), condom with spermicidal foam/gel/film/cream/suppository, diaphragm or cervical vault cap, or hormonal birth control (pills or injections). NOTE: Females are considered of childbearing potential unless they are surgically sterile (they have undergone a hysterectomy, bilateral tubal ligation, or bilateral oophorectomy) or they are postmenopausal (a woman who is ≥45 years of age and has not had menses for greater than 1 year).
9. Male subjects without a previous vasectomy should agree to use an adequate method of contraception (i.e. abstinence, condom with spermicidal foam/gel/film/cream) starting with the first dose of study therapy through 120 days after the last dose of study therapy.
10. Subjects with urothelial carcinoma must have received a prior platinum-based regimen in the metastatic setting or have signed consent for this study within 12 months of receiving a platinum-based regimen in the perioperative setting (neoadjuvant or adjuvant).
11. Subjects with a history of diabetes mellitus must have HgbA1c level of <8.5% upon study entry.

Subject Exclusion Criteria

The subject must be excluded from participating in the trial if the subject:

1. Is currently participating and receiving study therapy or has participated in a study of an investigational agent and received study therapy or used an investigational device within 4 weeks of the first dose of treatment.
2. Has a diagnosis of immunodeficiency or is receiving systemic steroid therapy or any other form of immunosuppressive therapy within 7 days prior to the first dose of trial treatment.
3. Has active TB (Bacillus Tuberculosis)
4. Hypersensitivity to pembrolizumab or any of its excipients.
5. Has had a prior anti-cancer monoclonal antibody (mAb) within 4 weeks prior to Cycle 1 Day 1 or who has not recovered (i.e. ≤ Grade 1 or at baseline) from adverse events due to agents administered more than 4 weeks earlier.
6. Has had prior chemotherapy, targeted small molecule therapy, or radiation therapy within 2 weeks prior to Cycle 1 Day 1 or who has not recovered (i.e. ≤ Grade 1 or at baseline) from adverse events due to a previously administered agent.

   * Note: Subjects with ≤ Grade 2 neuropathy are an exception to this criterion and may qualify for the study.
   * Note: If subject received major surgery, they must have recovered adequately from the toxicity and/or complications from the intervention prior to starting therapy.
7. Has a known additional malignancy that is progressing or requires active treatment. Exceptions include basal cell carcinoma of the skin or squamous cell carcinoma of the skin that has undergone potentially curative therapy or in situ cervical cancer.
8. Has known active central nervous system (CNS) metastases and/or carcinomatous meningitis. Subjects with previously treated brain metastases may participate provided they are stable (without evidence of progression by imaging for at least four weeks prior to the first dose of trial treatment and any neurologic symptoms have returned to baseline), have no evidence of new or enlarging brain metastases, and are not using steroids for at least 7 days prior to trial treatment. This exception does not include carcinomatous meningitis which is excluded regardless of clinical stability.
9. Has active autoimmune disease that has required systemic treatment in the past 2 years (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (e.g. thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment.
10. Has known history of, or any evidence of active, non-infectious pneumonitis.
11. Has an active infection requiring systemic therapy.
12. Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the subject's participation for the full duration of the trial, or is not in the best interest of the subject to participate, in the opinion of the treating investigator.
13. Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
14. Is pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the trial, starting with the pre-screening or screening visit through 120 days after the last dose of trial treatment.
15. Has received prior therapy with an anti-PD-1, anti-PD-L1, or anti-PD-L2 agent (only during Dose Expansion Phase Cohort A).
16. Has a known history of Human Immunodeficiency Virus (HIV) (HIV 1/2 antibodies).
17. Has known active Hepatitis B (e.g. HBsAg reactive) or Hepatitis C (e.g. HCV RNA [qualitative] is detected).
18. Has received a live vaccine within 30 days of planned start of study therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2016-02-23 (Actual); Primary Completion 2023-03-28 (Actual); Study Completion 2023-03-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Roberto Pili, MD, Principal Investigator — Indiana University School of Medicine, Indiana University Simon Cancer Center
Locations (4):
- United States (4):
  - USC/Norris Comprehensive Cancer Center, Los Angeles, California
  - Indiana University Hospital, Indianapolis, Indiana
  - Indiana University Melvin and Bren Simon Cancer Center, Indianapolis, Indiana
  - Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins, Baltimore, Maryland

REFERENCES:
- [Derived] Pili R, Quinn DI, Adra N, Logan T, Colligan S, Burney HN, Hahn NM. A Phase I/IB, Open Label, Dose Finding Study to Evaluate Safety, Pharmacodynamics and Efficacy of Pembrolizumab in Combination With Vorinostat in Patients With Advanced Prostate, Renal or Urothelial Carcinoma. Cancer Med. 2025 Apr;14(7):e70725. doi: 10.1002/cam4.70725. PMID 40145367

RESULTS

PARTICIPANT FLOW:
Groups:
- Dose Finding Cohort Dose Level 1: Patients were treated with 100 mg of oral vorinostat every day for 14 days, and with pembrolizumab at the fixed dose of 200 mg IV on day one of each cycle. Each cycle lasted 21 days. Patients had either previously treated, progressive renal or urothelial cell carcinoma that was locally advanced or metastatic, or progressive prostate cancer that was locally advanced or metastatic.
- Dose Finding Cohort Dose Level 2: Patients were treated with 200 mg of oral vorinostat every day for 14 days, and with pembrolizumab at the fixed dose of 200 mg IV on day one of each cycle. Each cycle lasted 21 days. Patients had either previously treated, progressive renal or urothelial cell carcinoma that was locally advanced or metastatic, or progressive prostate cancer that was locally advanced or metastatic.
- Expansion Cohort A: Patients with anti-PD1 naïve renal and urothelial cell carcinoma were treated with 200 mg of oral vorinostat every day for 14 days, and with pembrolizumab at the fixed dose of 200 mg IV on day one of each cycle. Each cycle lasted 21 days. Patients had to have previously undergone cancer treatment and have progressive disease that was locally advanced or metastatic.
- Expansion Cohort B: Patients with anti-PD1 resistant renal and urothelial cell carcinoma were treated with 200 mg of oral vorinostat every day for 14 days, and with pembrolizumab at the fixed dose of 200 mg IV on day one of each cycle. Each cycle lasted 21 days. Patients had to have previously undergone cancer treatment and have progressive disease that was locally advanced or metastatic.
- Expansion Cohort C: Patients with androgen-sensitive or castration-resistant prostate cancer were treated with 200 mg of oral vorinostat every day for 14 days, and with pembrolizumab at the fixed dose of 200 mg IV on day one of each cycle. Each cycle lasted 21 days. Patients had to have progressive disease that was locally advanced or metastatic.
Period: Overall Study
Arm/Group | Dose Finding Cohort Dose Level 1 | Dose Finding Cohort Dose Level 2 | Expansion Cohort A | Expansion Cohort B | Expansion Cohort C
Started | 4 | 4 | 15 | 14 | 15
Completed | 0 | 0 | 1 | 0 | 0
Not Completed | 4 | 4 | 14 | 14 | 15
Not completed — Adverse Event | 0 | 0 | 1 | 1 | 3
Not completed — Alternative Therapy | 0 | 0 | 1 | 0 | 0
Not completed — Death | 0 | 0 | 0 | 1 | 0
Not completed — Disease Progression | 4 | 2 | 8 | 9 | 10
Not completed — Needed a disqualifying therapy | 0 | 0 | 1 | 0 | 0
Not completed — Transferred to hospice | 0 | 0 | 1 | 0 | 0
Not completed — Physician Decision | 0 | 1 | 2 | 3 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 0 | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Dose Finding Cohort Dose Level 1 | Dose Finding Cohort Dose Level 2 | Expansion Cohort A | Expansion Cohort B | Expansion Cohort C | Total
Number analyzed (Participants) | 4 | 4 | 15 | 14 | 15 | 52
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 1 | 1 | 6 | 6 | 1 | 15
  >=65 years | 3 | 3 | 9 | 8 | 14 | 37
Age, Continuous [Mean (Standard Deviation); unit: years] | 66.2 (12.4) | 69.3 (7.8) | 64.3 (8.6) | 65.4 (10.3) | 69.0 (6.5) | 66.5 (8.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 2 | 3 | 4 | 0 | 11
  Male | 2 | 2 | 12 | 10 | 15 | 41
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 2 | 1 | 0 | 3
  Not Hispanic or Latino | 4 | 4 | 13 | 13 | 15 | 49
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 2 | 2
  White | 4 | 4 | 13 | 14 | 13 | 48
  More than one race | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 2 | 0 | 0 | 2
Region of Enrollment [Number; unit: participants]
  United States | 4 | 4 | 15 | 14 | 15 | 52
ECOG Performance Status [Count of Participants; unit: Participants] — 0. Fully active, able to carry on all pre-disease performance without restriction
  1. Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature, e.g., light house work, office work
  2. Ambulatory and capable of all selfcare but unable to carry out any work activities; up and about more than 50% of waking hours
  3. Capable of only limited selfcare; confined to bed or chair more than 50% of waking hours
  4. Completely disabled; cannot carry on any selfcare; totally confined to bed or chair
  5. Dead
  Participants
    0 | 1 | 1 | 6 | 4 | 4 | 16
    1 | 3 | 3 | 8 | 9 | 10 | 33
    2 | 0 | 0 | 1 | 0 | 1 | 2
    Missing | 0 | 0 | 0 | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate (Percentage of Patients With Complete Response or Partial Response)
Description: Measured by RECIST v1.1 Complete response: Disappearance of all target lesions Partial response: At least a 30% decrease in the sum of the longest diameter of target lesions, taking as reference the baseline sum longest diameter The percentage of patients with objective response and its 95% confidence interval will be provided.
Time Frame: Up to 4.5 years
Population: Patients were considered eligible for this analysis if they were in the expansion cohorts and had at least one follow-up assessment of disease status after completing one cycle of combination therapy.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Expansion Cohort A | Expansion Cohort B | Expansion Cohort C
Number analyzed (Participants) | 13 | 11 | 12
percentage of participants | 7.7 [0.2 to 36.0] | 0 [0 to 28.5] | 16.7 [2.1 to 48.4]

2. Primary Outcome: Progression Free Survival
Description: Progression free survival was determined from start date of treatment to date of progression for patients who progressed or date of death for patients who died without progressing. The observations of patients remaining alive and progression free were censored at the date of last disease evaluation. The Kaplan-Meier method was used to determine the median and 95% confidence interval.
Time Frame: Up to 4.5 years
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Expansion Cohort A | Expansion Cohort B | Expansion Cohort C
Number analyzed (Participants) | 13 | 11 | 12
months | 2.9 [1.3 to 21.8] | 3.5 [2.5 to 7.2] | 3.5 [1.3 to 7.5]

3. Secondary Outcome: Safety and Tolerablity: Number of Patients Who Experienced Grade 3 or 4 Adverse Events
Description: Number of unique patients who had a treatment-related (possible, probable, or definite) adverse event with grade 3 or greater using the Common Terminology Criteria for Adverse Events (CTCAE) version 4.0.
Time Frame: Up to 4.5 years
Population: Patients who received at least one dose of either study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Dose Finding Cohort Dose Level 1 | Dose Finding Cohort Dose Level 2 | Expansion Cohort A | Expansion Cohort B | Expansion Cohort C
Number analyzed (Participants) | 4 | 4 | 15 | 14 | 15
Participants | 0 | 0 | 5 | 3 | 5

4. Secondary Outcome: Number of Patients Experiencing a Dose Limiting Toxicity
Description: Dose limiting toxicities (DLTs) are defined as Grade ≥ 3 hematological/non hematological toxicities attributable to vorinostat and/or pembrolizumab during the first 21 days of the combination treatment (days 1-21). If DLTs occur in 1 patient treated at the starting dose level a minimum of another 3 patients will be treated at this dose level. If a DLT occurs in more than 1 patient in the first 6 patients the study will be terminated. If a DLT occurs in < 1/3 patients or ≤ 1/6 patients, 3 additional patients will be treated at the next dose level (level 2) with 200 mg vorinostat PO. If no DLTs occur at dose level 2, this dose level will be recommended for the expansion cohorts of the study.
Time Frame: Up to 21 days
Population: Patients who completed one cycle of study therapy.
Measure: Count of Participants; unit: Participants
Arm/Group | Dose Finding Cohort Dose Level 1 | Dose Finding Cohort Dose Level 2
Number analyzed (Participants) | 3 | 3
Participants | 0 | 0

ADVERSE EVENTS:
Time Frame: Up to 4.5 years
Arm/Group | Dose Finding Cohort Dose Level 1 | Dose Finding Cohort Dose Level 2 | Expansion Cohort A | Expansion Cohort B | Expansion Cohort C
All-Cause Mortality (participants affected / at risk) | 4/4 | 4/4 | 11/15 | 13/14 | 11/15
Serious Adverse Events (participants affected / at risk) | 3/4 | 2/4 | 10/15 | 6/14 | 5/15
Other Adverse Events (participants affected / at risk) | 4/4 | 4/4 | 15/15 | 13/14 | 14/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dose Finding Cohort Dose Level 1 (N=4) | Dose Finding Cohort Dose Level 2 (N=4) | Expansion Cohort A (N=15) | Expansion Cohort B (N=14) | Expansion Cohort C (N=15)
Anemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (3) | 1 (1) | 0 (0)
Death NOS (General disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
Nervous system disorders - Other (Nervous system disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Thromboembolic event (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Adult respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Blood bilirubin increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cardiac arrest (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Fever (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastrointestinal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hematuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hyperthyroidism (Endocrine disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyponatremia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypothyroidism (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ileus (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Joint infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Localized edema (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pain (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Renal and urinary disorders - Other (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Respiratory, thoracic and mediastinal disorders - Other (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Stroke (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dose Finding Cohort Dose Level 1 (N=4) | Dose Finding Cohort Dose Level 2 (N=4) | Expansion Cohort A (N=15) | Expansion Cohort B (N=14) | Expansion Cohort C (N=15)
Anemia (Blood and lymphatic system disorders) | 2 (4) | 2 (7) | 10 (16) | 2 (4) | 3 (8)
Fatigue (General disorders) | 2 (5) | 1 (3) | 11 (18) | 4 (6) | 6 (6)
Nausea (Gastrointestinal disorders) | 3 (4) | 1 (1) | 10 (14) | 6 (7) | 10 (10)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 3 (3) | 4 (12) | 2 (2) | 8 (14)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (3) | 8 (9) | 4 (6) | 4 (5)
Anorexia (Metabolism and nutrition disorders) | 3 (4) | 2 (2) | 7 (8) | 5 (6) | 4 (4)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 1 (3) | 7 (10) | 4 (5) | 3 (4)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 2 (21) | 2 (2) | 0 (0)
Vomiting (Gastrointestinal disorders) | 3 (4) | 2 (3) | 5 (7) | 3 (4) | 3 (3)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 7 (11) | 2 (3) | 4 (5)
Urinary tract infection (Infections and infestations) | 3 (5) | 0 (0) | 3 (8) | 1 (3) | 1 (1)
Creatinine increased (Investigations) | 0 (0) | 2 (3) | 3 (8) | 1 (2) | 1 (2)
Hyperglycemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 4 (15) | 0 (0) | 0 (0)
Pain (General disorders) | 1 (1) | 1 (1) | 2 (4) | 2 (3) | 3 (6)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 6 (6) | 1 (1) | 4 (5)
Hypophosphatemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 2 (3) | 1 (3) | 3 (7)
Fever (General disorders) | 1 (1) | 1 (1) | 3 (4) | 0 (0) | 3 (6)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 1 (6) | 1 (2) | 4 (4)
Edema limbs (General disorders) | 0 (0) | 0 (0) | 4 (6) | 1 (1) | 3 (3)
Hyperuricemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (7) | 1 (2) | 1 (1)
Hypothyroidism (Endocrine disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (4) | 5 (5)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 4 (8) | 1 (1) | 1 (1)
Insomnia (Psychiatric disorders) | 0 (0) | 0 (0) | 6 (8) | 0 (0) | 1 (1)
Alkaline phosphatase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (8)
Dehydration (Metabolism and nutrition disorders) | 1 (2) | 0 (0) | 3 (3) | 0 (0) | 3 (3)
Hyponatremia (Metabolism and nutrition disorders) | 1 (2) | 0 (0) | 3 (3) | 1 (1) | 2 (2)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 0 (0) | 3 (3) | 0 (0) | 1 (3)
Hyperkalemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 3 (6) | 1 (1) | 0 (0)
Platelet count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 2 (4)
Weight loss (Investigations) | 0 (0) | 1 (1) | 3 (4) | 2 (2) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0) | 3 (3) | 1 (1) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2) | 3 (4) | 0 (0)
Hypokalemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (2) | 3 (3) | 0 (0)
Hypotension (Vascular disorders) | 1 (1) | 1 (1) | 2 (2) | 1 (1) | 1 (1)
Upper respiratory infection (Infections and infestations) | 0 (0) | 0 (0) | 4 (4) | 1 (2) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 3 (3)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 1 (1)
Chills (General disorders) | 1 (1) | 0 (0) | 3 (3) | 0 (0) | 1 (1)
Dry mouth (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Dysgeusia (Nervous system disorders) | 1 (1) | 0 (0) | 2 (2) | 1 (1) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 2 (2)
Alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 1 (1)
Blurred vision (Eye disorders) | 0 (0) | 0 (0) | 2 (4) | 0 (0) | 0 (0)
Edema face (General disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 1 (1)
Flatulence (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (2)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 2 (2) | 1 (1) | 1 (1) | 0 (0)
Hypercalcemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 2 (2) | 0 (0) | 0 (0)
Papulopustular rash (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (4)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (3) | 1 (1) | 0 (0)
Skin and subcutaneous tissue disorders - Other (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 2 (2)
Skin infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (4) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3)
Anxiety (Psychiatric disorders) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Colitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 1 (1)
Conjunctivitis (Eye disorders) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Flu like symptoms (General disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 1 (1)
Fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Hypomagnesemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Peripheral sensory neuropathy (Nervous system disorders) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 0 (0)
Proteinuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Blood bilirubin increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Bruising (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Depression (Psychiatric disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ear pain (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Endocrine disorders - Other (Endocrine disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Hot flashes (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Hyperthyroidism (Endocrine disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypoalbuminemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Infusion related reaction (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Non-cardiac chest pain (General disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Pelvic pain (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Penile pain (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Rash acneiform (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Soft tissue infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Urinary frequency (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Agitation (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Allergic reaction (Immune system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anal fistula (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Anal hemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ataxia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bladder infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Bloating (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Breast pain (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cardiac troponin I increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chest wall pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cholesterol high (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dry eye (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Duodenal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Eye disorders - Other (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastrointestinal disorders - Other (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastrointestinal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Heart failure (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hematoma (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hematuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hemorrhoids (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Flank pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypocalcemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypoglycemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Infections and infestations - Other (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Injury, poisoning and procedural complications - Other (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Investigations - Other (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Leukocytosis (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lip infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lower gastrointestinal hemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lung infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lymphocyte count decreased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Memory impairment (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Movements involuntary (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Mucositis oral (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Muscle weakness trunk (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal and connective tissue disorder - Other (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nail discoloration (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nervous system disorders - Other (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Oral pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Palmar-plantar erythrodysesthesia syndrome (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Paresthesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Penile infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Peritoneal infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Presyncope (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Respiratory, thoracic and mediastinal disorders - Other (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sinus disorder (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Skin induration (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Skin ulceration (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Stomach pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Toothache (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Urinary retention (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Wound dehiscence (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Wound infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-04-07): https://cdn.clinicaltrials.gov/large-docs/53/NCT02619253/Prot_SAP_000.pdf